CLINICAL TRIAL: NCT02294136
Title: Intervention to Improve HCV Treatment Uptake and Adherence in HIV/HCV Coinfection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GCO 12-0693; R34MH099930-02 (NIH)
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: HIV; Hepatitis C; Co-Infection
Keywords: HIV; HCV; Adherence; Psychiatric; Behavioral; Intervention
MeSH Terms: conditions — Hepatitis C; Coinfection; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prep-C (Experimental): Four session nurse administered behavioral intervention.
  Interventions: Behavioral: Prep-C
- Educational Control (Active Comparator): Attention Control
  Interventions: Behavioral: Educational Control

INTERVENTIONS:
Behavioral: Prep-C — PREP-C is a web-based structured clinical interview that healthcare providers of diverse disciplines can be trained to administer. It provides an assessment of a client's psychosocial readiness to begin HCV treatment and identifies domains of functioning which require tailored intervention to improve treatment readiness.
  Arms: Prep-C
Behavioral: Educational Control — Attention Control
  Arms: Educational Control

SUMMARY:
End-stage liver disease, predominantly due to hepatitis C virus (HCV) infection, is one of the leading causes of death in person living with HIV infection. While HCV is curable and recent advances in treatment have increased the rates of cure, few patients with HIV and HCV are being treated to cure HCV. Based on formative research, the investigators developed the "Psychosocial Readiness Evaluation and Preparation for hepatitis C treatment (PREP-C)". PREP-C is a clinical interview that healthcare providers of diverse disciplines can be trained to administer. It provides an assessment of a client's psychosocial readiness to begin HCV treatment and identifies domains of functioning which require intervention to improve treatment readiness. PREP-C (www.prepC.org) is also a telemedicine resource for health care providers. Under this protocol, the existing PREP-C clinical interview (or assessment) is incorporated with a behavioral intervention. This study tests the integrated assessment-behavioral intervention to increase HCV treatment initiation among HIV-co-infected patients. The assessment-behavioral intervention under this protocol is conducted in two phases, an Intervention Development phase and a Pilot Randomized Clinical Trial (RCT) phase.

Findings from this vanguard study will inform the design parameters of a larger, more rigorous evaluation in an R01 application, if results are promising. The PREP-C web-based assessment and intervention package is designed to be scalable and can be disseminated through the live PrepC.org web site. The proposed study is innovative in that it seeks to develop the first web-based intervention for health care providers to use to increase HCV treatment initiation in HIV/HCV-co-infected persons. The study can have a major public health impact by providing needed structured resources for health care providers to increase rates of HCV treatment initiation in HIV/HCV-co-infected persons, thereby reducing mortality due to end-stage liver disease.

DETAILED DESCRIPTION:
In response to PAR-12-279 "Pilot Intervention and Services Research Grants (R34)," this application proposes to develop and to test the feasibility, acceptability, and preliminary efficacy of a nurse-delivered intervention addressing patient-level barriers (Information, Motivation, and Behavioral Skills) to hepatitis C virus (HCV) treatment uptake and adherence in HIV-co-infected patients. End-stage liver disease is a leading cause of mortality in HIV-infected persons as a result of high rates of untreated chronic HCV-co-infection. HCV infection can be cured and the effectiveness of HCV treatment has dramatically increased with the FDA approval of two HCV protease inhibitors in May 2011. The uptake of HCV treatment in HIV/HCV-co-infected patients remains, however, unacceptably low (estimated at 10%) despite the fact that testing has been standard of care for all HIV-infected persons for over 10 years. Progress in developing effective behavioral interventions to successfully engage and retain HIV-co-infected patients who are already engaged in HIV care in HCV care has not kept pace with the significant pharmacologic advances in HCV treatment.

There are multiple barriers to HCV treatment initiation at patient, provider, and structural levels. As HCV treatment becomes more effective and more clinics overcome the structural and provider barriers, there will be an increasing need for a structured means to assess patient-level barriers and provide effective interventions in order to increase HCV treatment initiation, adherence, and cure rates in HIV/HCV-co-infected patients.

Based on formative prior NIH research (K23MH71177), the investigators have developed the "Psychosocial Readiness Evaluation and Preparation for hepatitis C treatment (PREP-C)". PREP-C is a web-based structured clinical interview that healthcare providers of diverse disciplines can be trained to administer. It provides an assessment of a client's psychosocial readiness to begin HCV treatment and identifies domains of functioning which require tailored intervention to improve treatment readiness. PREP-C has to date been administered by the PI (Weiss) to 97 patients and a telemedicine resource for health care providers was launched in July 2012 (PrepC.org).

Specific aims:

1. To formally adapt existing behavioral medicine interventions based on PREP-C assessment to target individual barriers (Information, Motivation, and Behavior Skills) to HCV treatment initiation in HIV/HCV-co-infected patients who are medically eligible for HCV treatment, pilot test and refine the tailored intervention in 15 HIV/HCV-co-infected patients, and finalize the intervention manual.
2. To conduct a pilot randomized clinical trial with 60 HIV/HCV-co-infected patients who are medically eligible for HCV treatment, comparing the nurse-delivered PREP-C intervention (n=30) with attention control (n=30) in order to evaluate patient acceptance, patient satisfaction, enrollment and retention, as well as preliminary efficacy (initiation of HCV treatment within 6 months of randomization and persistence and adherence to the first 12 weeks of treatment in those who do initiate treatment).

Hypothesis: The PREP-C intervention will increase Motivation, Information, and Self-Efficacy leading to higher rates of HCV treatment initiation, persistence and adherence in the PREP-C intervention arm.

The intervention to be studied is guided by the Information-Motivation-Behavioral Skills Model of health behavior to adapt Motivational Interviewing and Cognitive-Behavioral Therapy techniques (e.g., cognitive restructuring) to the specific needs of this patient population. In this study, a nurse will be trained to administer the PREP-C integrated assessment-behavioral intervention. This four-session integrated assessment-intervention includes administration of already developed PREP-C assessment in session one, and tailored interventions targeting Motivation, Information and Behavioral Skills in sessions 2-4 to be developed in this study. The research will take place at a major academic medical center in which HIV/HCV-co-infected patients are actively being treated for HCV infection.

Findings from this vanguard study will inform the design parameters of a larger, more rigorous evaluation in an R01 application, if results are promising. The PREP-C web-based assessment and intervention package is designed to be scalable and can be disseminated through the live PrepC.org web site. The proposed study is innovative in that it seeks to develop the first web-based intervention for health care providers to use to increase HCV treatment initiation in HIV/HCV-co-infected persons. The study can have a major public health impact by providing needed structured resources for health care providers to increase rates of HCV treatment initiation in HIV/HCV-co-infected persons, thereby reducing mortality due to end-stage liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Co-infected with HIV and HCV
* 21 years and older
* Primary language is English or Spanish
* Two most recent HIV RNA levels are both <1000 copies/mL
* Has attended appointment with HIV PCP in previous 6 months
* Has not attended appointment with HCV Provider in last year

Exclusion Criteria:

* Presence of active malignancy (except for squamous or basal cell skin cancers), not otherwise in remission
* Chronic kidney disease in hemodialysis or peritoneal dialysis
* Decompensated cirrhosis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-12; Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Hepatitis C Treatment Initiation | 6 months post intervention
  Whether or not subject has initiated Hepatitis C treatment within 6 months of study randomization.

SECONDARY OUTCOMES:
Adherence to Hepatitis C Treatment | up to 6 months
  Adherence to Hepatitis C medications will be assessed for subjects who initiate Hepatitis C treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Weiss, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States